CLINICAL TRIAL: NCT01474265
Title: Alterations in the Autonomic Nervous System During Smoking Quit Attempts- Possible Effects of Pharmacological Interventions
Brief Title: Sympathovagal Balance in Smoking Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Collaborators: University Medical Center Goettingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201102-TR
Record Dates: First submitted 2011-11-03; First posted 2011-11-18 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; varenicline; sympathovagal balance; quit attempts; MSNA
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- varenicline placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- varenicline (Active Comparator)
  Interventions: Drug: Varenicline
- Nicorette TX (Active Comparator)
  Interventions: Drug: Nicorette TX
- Nicorette TX optional (Active Comparator)
  Interventions: Drug: Nicorette TX
- control group smokers (No Intervention)

INTERVENTIONS:
Drug: Varenicline — 0.5-2 mg per day, oral use
  Arms: varenicline
Drug: Placebo — 1-2 tablets per day, oral use
  Arms: varenicline placebo
Drug: Nicorette TX — 10-15 mg per day, transdermal use (patches)
  Arms: Nicorette TX; Nicorette TX optional

SUMMARY:
This study has the following primary aim:

- the main objective of this study is to investigate the effects of smoking cessation during quit attempts on sympathovagal balance. These effects will be observed in smokers quitting smoking with pharmacological support or without.

Secondary aims of this study are also:

* the definition of MSNA in smokers and non-smokers
* the investigation of other parameters concerning the autonomic nervous system, like baroreflex-sensitivity, heart rate-variability before and during the quit attempt.
* the definition of withdrawal symptoms and craving before, during and after the quit attempt.
* the investigation of effects of smoking cues on craving and sympathovagal balance
* the investigation of relapse rates after smoking cessation in correlation with the parameters mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women at the age of 25 to 60 years.
* Group A-D: Smokers willing to quit smoking and a FTNA-result >5.
* Group E: Never-smokers.
* Signed consent after information.

Exclusion Criteria:

* formerly known hypersensitivity against one of the used pharmacological interventions or structurally similar drugs or against one of the ingredients.
* participation in another study during this study or within 4 weeks prior to this study.
* Addiction or other circumstances that prevent the patient from estimating the study and the consequences.
* Pregnancy and breast-feeding
* women with childbearing potential, except women that fulfill the following criteria:

  * post menopause
  * postoperative (6 weeks after both-sides ovariectomy with or without hysterectomy)
  * regular and correct use of prevention methods (error-rate <1% a year), e.g. implants, depot injections, oral contraceptives, IUP)
  * sexual abstinence
* signs that predict a possible non-compliance of the patient
* exclusion because of nicorette tx:

  * psoriasis, dermatitis, urticaria
* exclusion because of varenicline

  * creatinine-clearance < 30ml/min
  * epilepsy
  * psychiatric diseases (schizophrenia, bipolar disorders, depression).
* Exclusion because of methods

  * Diseases that increase the sympathetic level (Heart insufficiency, high blood pressure (arteria /pulmonary), obstructive sleeping apnoea, COPD)
* cardiac rhythm disturbances
* myocardial infarction within the last 8 weeks
* polyneuropathy
* diseases that come along with damages of peripheral nerves
* severe or life-threatening diseases (e.g. cancer with life-expectancy < 5 years, terminal kidney-insufficiency)
* treatment with antihypertensive drugs or sympathomimetic substances (e.g.theophyllin) or smoking cessation medication (NRT, Varenicline)
* Other reasons, that make a patient not suitable for the study (estimation of primary investigator)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Assessment of muscular sympathic nervous activity (MSNA) in bursts / 100 heart beats before and while smoking cessation. | 33 weeks
  Patients present 7 weeks before their personal smoking-stop-day and participate in the study until week 26 after their personal smoking-stop-day. During that time, MSNA is recorded.

SECONDARY OUTCOMES:
Assessment of the basal sympathetic nerve activity in smokers compared to never-smokers | 33 weeks
  first MSNA is carried out 4 weeks before smoking-stop-day (respectively 6 weeks for group D). second and last MSNA is carried out two days after smoking-stop-day (respectively 2 weeks before smoking-stop-day for group D)
Assessment of craving and withdrawal symptoms during smoking cessation | 33 weeks
  withdrawal symptoms data is collected by phone calls 3,2,1 days before smoking-stop-day, the day itself and 1 day and 11 (12 for group C and D) weeks after smoking-stop-day.
  Also the withdrawal symptoms date is collected during each personal examination (means - Pre-Examination, Baseline, Follow I to III).
  The data will be collected by reliable questionnaires
Assessment of smoking cues on craving and sympathovagal balance | 33 weeks
  smoking cues will be presented on the first follow-up-measurement to members of group A-D.
Assessment of smoking relapse rate | 33 weeks
  All relapses will be registered to correlate them with the obtained parameters (baroreflex-sensitivity, heartrate-variabilty, MSNA, questionnaires)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Raupach, MD, Principal Investigator — University Medical Center Goettingen
Locations (1):
- University Medical Center, Göttingen, Germany